CLINICAL TRIAL: NCT04351373
Title: Microscopic Fluorescence-guided Vestibular Schwannoma, Meningioma, Head and Neck Paraganglioma, or Head and Neck Schwannoma Resection Using Fluorescein Sodium and YELLOW 560
Brief Title: Microscopic Fluorescence-guided Vestibular Schwannoma Resection Using Fluorescein Sodium and YELLOW 560
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Matthew L. Carlson, M.D., Principal Investigator, Mayo Clinic
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 19-005178
Record Dates: First submitted 2020-04-09; First posted 2020-04-17 (Actual); Results first posted 2023-08-01 (Actual); Last update posted 2023-08-01 (Actual); Status verified 2023-07

CONDITIONS: Vestibular Schwannoma
Keywords: Head and Neck Paraganglioma; Head and Neck Schwannoma
MeSH Terms: conditions — Neuroma, Acoustic | interventions — Fluorescein; Fluoresceins

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: Yes

ARMS (1):
- Fluorescein sodium (FS) and YELLOW 560 nm microscope filter (YE560) during surgery (Experimental): Subjects undergoing clinically planned vestibular schwannoma, Meningioma, Head and Neck Paraganglioma, or Head and Neck Schwannoma, removal surgery will have contrast agent fluorescein sodium administered intravenously after tumor exposure, and a special filter called YELLOW560 will be used on the operating microscope to see the fluorescent coloring of the contrast.
  Interventions: Drug: Fluorescein Sodium; Device: YELLOW560 filter

INTERVENTIONS:
Drug: Fluorescein Sodium — Intravenous administration 1 mg/kg initial dosing if insufficient additional doses of 1 mg/kg may be administered.
  Other Names: AK-Fluor®
Device: YELLOW560 filter — Integrated fluorescence module serves to make fluorescent areas visible to assist in visualizing tumor during the resection.
  Other Names: YELLOW 560 nm microscope filter (YE560)

SUMMARY:
The purpose of this study is to see if there is benefit to using an IV contrast called AK-Fluor® and a microscope filter called YELLOW560 when surgically removing a vestibular schwannoma, Meningioma, Head and Neck Paraganglioma, or Head and Neck Schwannoma.

ELIGIBILITY:
Inclusion Criteria

* Patient with a suspected VS
* Recurrent VS with prior microsurgical resection or radiation therapy
* Clinical indication for microsurgical resection

Exclusion Criteria

* History of allergy to FS
* History of renal failure
* Pregnant women
* Those with inability to give informed consent
* Prisoners and inmates

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2021-10-06 (Actual); Primary Completion 2022-05-25 (Actual); Study Completion 2022-05-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Matthew L Carlson, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Chan SA, Macielak RJ, Tuchscherer AM, Neff BA, Driscoll CLW, Peris-Celda M, Van Gompel JJ, Link MJ, Carlson ML. Fluorescein-Assisted Microsurgical Resection of Vestibular Schwannoma: A Prospective Feasibility Study. Otol Neurotol. 2022 Dec 1;43(10):1240-1244. doi: 10.1097/MAO.0000000000003718. Epub 2022 Oct 14. PMID 36240730
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Fluorescein Sodium (FS) and YELLOW 560 nm Microscope Filter (YE560) During Surgery
Started | 12
Completed | 11
Not Completed | 1
Not completed — Intraoperative diagnosis of facial nerve schwannoma | 1

BASELINE CHARACTERISTICS:
Arm/Group | Fluorescein Sodium (FS) and YELLOW 560 nm Microscope Filter (YE560) During Surgery
Number analyzed (Participants) | 12
Age, Continuous [Mean (Standard Deviation); unit: years] | 48 (15.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9
  Male | 3
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 12
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 12
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 12

OUTCOME MEASURES:

1. Primary Outcome: Surgeon Predicted Use of Fluorescein Sodium in Future Cases
Description: Physician response to surgeon survey question, "Based on the use and performance of FS in this case alone, how likely are you to use FS in future cases (excluding the research trial) involving this tumor?" using a Likert-style rating from 0-4 where 0=Unsure; 1= Plan to not use in any cases; 2= Plan to use in select cases; 3=Plan to use in the majority of cases; 4=Plan to use in all cases.
Time Frame: Approximately 3 months postoperatively
Measure: Number; unit: participants
Arm/Group | Fluorescein Sodium (FS) and YELLOW 560 nm Microscope Filter (YE560) During Surgery
Number analyzed (Participants) | 8
participants
  Unsure | 0
  Plan to not use in any cases | 0
  Plan to use in select cases | 4
  Plan to use in the majority of cases | 3
  Plan to use in all cases | 1

2. Primary Outcome: Correlation of Fluorescein Sodium With Surgeons' Visual Assessment
Description: Fluorescence correlate with surgeons' visual assessment of the tumor and nerve tissue under normal microscopy without the Yellow 560 filter using a Likert-style rating from 1-4 where 1=No correlation; 2=Some correlation; 3=Good correlation; 4=Excellent correlation.
Time Frame: Intraoperatively, approximately 1 day
Measure: Number; unit: participants
Arm/Group | Fluorescein Sodium (FS) and YELLOW 560 nm Microscope Filter (YE560) During Surgery
Number analyzed (Participants) | 8
participants
  No correlation | 1
  Some correlation | 0
  Good correlation | 1
  Excellent correlation | 6

3. Primary Outcome: Correlation of Fluorescein Sodium With Electrostimulation
Description: Surgeons' assessment of fluorescence correlate with electrostimulation (e.g. tissues with high fluorescence do not stimulate, whereas nerve tissues with low fluorescence do stimulate)" using a Likert-style rating from 1-4 where 1=No correlation; 2=Some correlation; 3=Good correlation; 4=Excellent correlation.
Time Frame: Intraoperatively, approximately 1 day
Measure: Number; unit: participants
Arm/Group | Fluorescein Sodium (FS) and YELLOW 560 nm Microscope Filter (YE560) During Surgery
Number analyzed (Participants) | 8
participants
  No correlation | 1
  Some correlation | 0
  Good correlation | 3
  Excellent correlation | 4

4. Secondary Outcome: Time to Differential Visualization
Description: The amount of time in minutes for differential visualization of the tumor and surrounding tissue after sodium fluorescein administration during surgery
Time Frame: Intraoperatively, approximately 1 day
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Fluorescein Sodium (FS) and YELLOW 560 nm Microscope Filter (YE560) During Surgery
Number analyzed (Participants) | 11
minutes | 41 (24)

5. Secondary Outcome: Average Dose of Sodium Fluorescein Administration
Description: Average dose of sodium fluorescein administered during surgery to achieve differential fluorescence of the tumor and tissue reported in mg/kg
Time Frame: Intraoperatively, approximately 1 day
Measure: Mean (Standard Deviation); unit: mg/kg
Arm/Group | Fluorescein Sodium (FS) and YELLOW 560 nm Microscope Filter (YE560) During Surgery
Number analyzed (Participants) | 11
mg/kg | 3.3 (0.8)

6. Secondary Outcome: Total Resection Rate
Description: Number of subjects to have a gross total resection
Time Frame: Intraoperatively, approximately 1 day
Measure: Count of Participants; unit: Participants
Arm/Group | Fluorescein Sodium (FS) and YELLOW 560 nm Microscope Filter (YE560) During Surgery
Number analyzed (Participants) | 11
Participants | 6

ADVERSE EVENTS:
Time Frame: Adverse events were collected from baseline to end of study participation for a total of approximately three months on all participants.
Arm/Group | Fluorescein Sodium (FS) and YELLOW 560 nm Microscope Filter (YE560) During Surgery
All-Cause Mortality (participants affected / at risk) | 0/12
Serious Adverse Events (participants affected / at risk) | 0/12
Other Adverse Events (participants affected / at risk) | 1/12
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Fluorescein Sodium (FS) and YELLOW 560 nm Microscope Filter (YE560) During Surgery (N=12)
Fever (General disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol (2021-11-25): https://cdn.clinicaltrials.gov/large-docs/73/NCT04351373/Prot_000.pdf